CLINICAL TRIAL: NCT07402798
Title: Respiration-induced Ablation Catheter Displacement and Anesthetic Safety of High-Frequency, Very-Low Tidal Volume Ventilation With Controlled Peak Pressure During Atrial Fibrillation Ablation: An Observational Crossover Pilot Study
Brief Title: Anesthetic Safety of High-Frequency, Very-Low Tidal Volume Ventilation With Controlled Peak Pressure During Atrial Fibrillation Ablation
Acronym: HFvLTVcPPSAFE
Status: Completed | Type: Observational
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Carlos Ramírez-Paesano,MD,PhD, Centro Medico Teknon
Other Study IDs: ICOR-25-HFvLTV; TKN-Ethical Committee (Other: TKNICOR_HFuLTV-cPP.2025)
Record Dates: First submitted 2026-01-26; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation (AF); Cardiac Arrhythmias
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, observational, within-subject crossover pilot study evaluates the impact of a high-frequency, very-low tidal volume ventilation strategy with controlled peak inspiratory pressure (HFvLTV-cPP) on respiration-induced ablation catheter displacement during atrial fibrillation (AF) radiofrequency ablation performed under general anesthesia. In the same patients, standard mechanical ventilation is compared with HFvLTV-cPP during the ablation phase to quantify catheter stability under matched contact force conditions. Secondary objectives include assessment of arterial carbon dioxide levels, ventilatory mechanics, hemodynamic parameters, anesthetic requirements, and post-anesthesia recovery outcomes. The study aims to determine whether limiting peak inspiratory pressure while using high respiratory rates and ultra-low tidal volumes improves catheter stability while maintaining acceptable gas exchange, cardiopulmonary safety, and postoperative recovery profiles.

DETAILED DESCRIPTION:
Catheter ablation is an established treatment for symptomatic atrial fibrillation (AF); however, recurrence after radiofrequency ablation remains frequent, with 30-40% of patients experiencing arrhythmia recurrence after a first procedure. Effective lesion formation depends on adequate catheter-tissue contact force and stability. General anesthesia improves catheter contact compared with conscious sedation by reducing thoracic motion, yet standard mechanical ventilation does not fully eliminate respiration-induced catheter displacement.

High-frequency jet ventilation has been shown to improve catheter stability but requires specialized equipment. As an alternative, high-frequency low tidal volume ventilation (HFLTV) using conventional anesthesia ventilators has been associated with reduced thoracic motion, improved catheter stability, and shorter ablation times. Nevertheless, sustained high respiratory rates may increase intrinsic positive end-expiratory pressure (PEEP), mechanical power, intrathoracic pressure, and carbon dioxide retention, and the safety profile of these strategies has not been fully characterized.

In addition, when tidal volume approaches anatomic and circuit dead space, effective alveolar ventilation decreases and PaCO₂ may rise, while increasing respiratory rate disproportionately increases mechanical power delivered to the respiratory system. Explicit limitation of peak inspiratory pressure, a factor rarely addressed in previous studies, may reduce ventilatory energy transfer, minimize catheter motion, and mitigate adverse cardiopulmonary effects.

High-frequency very-low tidal volume ventilation with controlled peak inspiratory pressure (HFvLTV-cPP) combines ultra-low tidal volumes with strict limitation of peak inspiratory pressure (≤ 20 cmH₂O) to minimize respiration-induced catheter displacement while preserving gas exchange, limiting mechanical power, and maintaining hemodynamic stability, accepting brief and controlled permissive hypercapnia.

Since 2021, HFLTV has been routinely implemented during AF ablation at the Instituto del Corazón (ICOR), Centro Médico Teknon (Barcelona, Spain). However, no prior studies have systematically evaluated a protocol incorporating explicit peak inspiratory pressure control, nor have they comprehensively assessed anesthetic recovery and post-anesthesia safety outcomes.

This prospective, observational, within-subject crossover pilot study was designed to compare standard mechanical ventilation with HFvLTV-cPP in the same patients undergoing radiofrequency catheter ablation for AF under general anesthesia. A one-way crossover design was used for ethical reasons, as HFLTV represents the institutional standard during the ablation phase. The study focuses on paired physiological and procedural differences rather than causal inference.

Adult patients (21-85 years) with paroxysmal, persistent, or permanent AF scheduled for radiofrequency ablation were enrolled. Exclusion criteria included severe ventricular dysfunction, significant valvular disease, severe pulmonary disease with auto-PEEP, pulmonary hypertension, uncontrolled asthma, chronic metabolic acidosis, and significant neurological disorders.

All procedures were performed under total intravenous anesthesia with propofol and remifentanil, with neuromuscular blockade and invasive arterial pressure monitoring. Mechanical ventilation was delivered using a standard anesthesia workstation, with tidal volumes calculated based on adjusted body weight.

Two ventilation strategies were applied sequentially in each patient:

Standard ventilation (baseline condition): tidal volume 6 mL/kg (adjusted body weight), respiratory rate 12 breaths/min, I:E ratio 1:2, FiO₂ 0.5, PEEP 0 cmH₂O.

HFvLTV-cPP during radiofrequency ablation: respiratory rate 50 breaths/min, I:E ratio 1:1, progressive reduction of tidal volume to ≤ 3 mL/kg (adjusted body weight) while maintaining peak inspiratory pressure ≤ 20 cmH₂O.

Ventilatory transitions were performed in a standardized stepwise manner, and measurements were obtained after physiological stabilization during each phase.

The primary outcome was respiration-related ablation catheter displacement, quantitatively measured (mm) at the same left atrial site under matched contact force (10 g) during standard ventilation and HFvLTV-cPP, and qualitatively assessed by the electrophysiologist.

Secondary outcomes included within-patient comparisons of arterial PaCO₂, ventilatory mechanics, hemodynamic variables, anesthetic and vasopressor requirements, procedural parameters, and post-anesthesia recovery outcomes. Postoperative recovery was evaluated using time to eye opening, time to extubation, Aldrete score, Richmond Agitation-Sedation Scale (RASS), and the incidence of respiratory or neurological complications.

Statistical analyses were limited to paired, within-subject comparisons using appropriate parametric or non-parametric tests. The study was designed as a pilot investigation to describe physiological, procedural, and recovery profiles associated with HFvLTV-cPP compared with standard ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21-85 years.
* Diagnosed with paroxysmal, persistent, or permanent atrial fibrillation (AF).
* Scheduled for radiofrequency ablation (RFA) under general anesthesia.
* Patients undergoing repeat ablation procedures included for evaluation of ventilatory, anesthetic, and post-anesthesia recovery parameters.
* Patients undergoing repeat ablation procedures excluded from analyses related to procedural efficacy outcomes.

Exclusion Criteria:

* Left or right ventricular dysfunction.
* Severe tricuspid regurgitation.
* Severe pulmonary hypertension.
* Severe chronic obstructive pulmonary disease (COPD) with evidence of auto-positive end-expiratory pressure.
* Uncontrolled severe asthma.
* Chronic metabolic acidosis with associated hyperkalemia.
* Severe migraine disorders.
* Trigeminal neuralgia.
* Atypical facial pain.
* Advanced hydrocephalus.
* Presence of ventriculoperitoneal shunt.
* Parkinson's disease.
* Epilepsy.
* Vertigo.
* Ménière's disease.
* Narrow-angle glaucoma.
* Prior stroke with persistent neurological deficits.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with paroxysmal, persistent, or permanent atrial fibrillation (AF) scheduled for radiofrequency ablation (RFA) under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-02-04 (Actual)

PRIMARY OUTCOMES:
Respiration related catheter stability during radiofrequency ablation. | Outcome measures were assessed intraprocedurally. Enrollement period was from May 2025 to September 2025.
  Respiration-related catheter stability was assessed quantitatively as catheter displacement (millimeters) during radiofrequency ablation. Catheter displacement was measured under standard mechanical ventilation and after 15 minutes of high-frequency, very low-tidal-volume ventilation with continuous positive pressure (HFvLTV-cPP).

CONTACTS AND LOCATIONS:
Locations (1):
- Teknon Medical Center, Barcelona, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided